CLINICAL TRIAL: NCT05645289
Title: Efficacy and Safety of Minodronate in the Treatment of Postmenopausal Osteoporosis With Low Back Pain: a Single-centre and Randomized Controlled Trial
Brief Title: Efficacy and Safety of Minodronate in Patients With Low Back Pain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M2022465
Record Dates: First submitted 2022-11-18; First posted 2022-12-09 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-11

CONDITIONS: Postmenopausal Osteoporosis
Keywords: minodronate; low back pain; adverse reactions; pharmacokinetic; pharmacodynamic
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Low Back Pain | interventions — YM 529; Alendronate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- minodronate (Experimental): Patients will take 1 mg of minodronate tablets orally in the morning.
  Interventions: Drug: Minodronate
- alendronate (Active Comparator): Patients will be orally given 10 mg alendronate tablets daily in the morning.
  Interventions: Drug: Alendronate

INTERVENTIONS:
Drug: Minodronate — The minodronate group: The group will include thirty-six patients. Patients will take 1 mg of minodronate tablets orally with 200 mL of water in the morning. They can not lie flat for at least 30 minutes after taking the tablets, and they can not eat anything except water for at least 30 minutes after taking the tablets once a day for 12 weeks, for a total of 84 times.
  Other Names: Difumi
  Arms: minodronate
Drug: Alendronate — The alendronate group: A total of 36 patients will be treated with alendronate. Patients will be orally given 10-mg alendronate tablets daily and 200 mL of water in the morning. They could not lie down and eat anything except water for at least 30 minutes after taking the tablets. The treatment lasted for 12 weeks, corresponding to a total of 84 doses.
  Other Names: Fushanmei
  Arms: alendronate

SUMMARY:
This study will provide objective evidence for the efficiency and safety of minodronate in the treatment of postmenopausal osteoporosis with low back pain protocol. Furthermore, it will be helpful to evaluate the quantitative relationship between bone metabolic markers (BTM) and bone mineral density (BMD) in patients with osteoporosis under different ages.

DETAILED DESCRIPTION:
The study is a randomized, parallel controlled clinical trial in Chinese postmenopausal OP patients receiving minodronate or alendronate. Minodronate will be administered once daily for 12 weeks, and alendronate will be administered once daily for 12 weeks. This study is divided into two stages: the first stage is 12 weeks, and at the end of the first stage, the results of patients' back pain and gastrointestinal adverse reactions will be summarized; the second stage is 12 weeks, and the pharmacokinetic and pharmacodynamic characteristics of patients will be summarized at the end of the second stage. The VAS score in this study rangs from 0-100 mm. During the screening, the patient's past pain relief methods, such as pain medication or the way of life intervention will be recorded. The use of the above methods during the patients' treatment will be prohibited to prevent interference with the results of the clinical trials. During the treatment, if patients experience sudden aggravation of low back pain, the VAS score is more than 70, and the patients could not bear the pain, a rescue drug (acetaminophen) will be used uniformly to relieve the pain. Throughout the trial, a total of 5 follow-up visits will be planned. The VAS score, PK&PD sampling, BMD evaluation, and Izumo scale score will be calculated.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese postmenopausal patients with a diagnosis of OP;
2. Patients with low back pain of at least 3 months and a VAS score ≥30;
3. The value of lumbar L1-4 or total hip bone density measured by DXA is < -2.5;
4. Serum 25-hydroxyvitamin D (25-OHD) concentration ≥20 ng/mL;
5. Patients with full capacity for civil conduct and understanding of the research process and methods voluntarily participated in this study and signed the informed consent form.

Exclusion Criteria:

1. Patient who are allergic to minodronate, alendronate, or other bisphosphonate drug or any other component of the drug under evaluation;
2. Patients with a diagnosis of secondary OP;
3. The following drugs affecting bone metabolism were used before the screening:

   Received injections of bisphosphonate and denosumab within 3 years; Received oral bisphosphonate, parathyroid hormones or analogues, strontium, or fluoride within 6 months; Received glucocorticoids, steroids, immunosuppressants, calcitonin, calcitriol or its analogues, thiazide diuretics, and ng-acting oestrogen/progesterone replacement therapy within 3 months;
4. Patients with a diagnosis of diseases affecting bone metabolism (e.g., osteogenesis imperfecta, malignancy, progressive diaphyseal dysplasia, Paget's disease, rheumatoid arthritis, osteosclerosis, osteoporosis with a slipped disc and spinal stenosis, and liver and kidney failure);
5. Patients are participating or have participated in an investigational drug study within 3 months before signing the informed consent form;
6. Patients under 75 years old with a creatinine clearance rate < 60 mL/min and those > 75 years old with a creatinine clearance rate < 45 mL/min;
7. Serum calcium levels < 2.0 mmol/L (8 mg/dL) or > 2.7 mmol/L (11.0 mg/dL);
8. Patients with fever, severe infection, severe trauma, or major surgery within 30 days;
9. Patients with a QTc interval of > 480 ms;
10. Patients are undergoing or planning to undergo invasive dental treatment;
11. Smoking history in the past six months;
12. Patients with a history of alcohol abuse (> 15 g of alcohol per day, equivalent to 350 mL of beer or 150 mL of wine, more than twice per week) and drug abuse;
13. Patients with a prior history of cerebral infarction, ischaemic or haemorrhagic stroke;
14. Patients with implants and/or fractures in the lumbar spine or hip that interfere with BMD testing;
15. Received pain relievers (e.g., nonsteroidal anti-inflammatory drugs, central analgesics) or life interventions to relieve pain within 1 week before screening;

Ages: 55 Years to 95 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
The time for a 10 point decrease in the VAS score within 24 weeks | up to 24 weeks
  The VAS scores were measured daily within 24 weeks. Back pain was evaluated using a 100-mm VAS score ( 0 = no pain, 100 = worst pain possible) after treatment, where the patients recorded their pain on the VAS by themselves everyday.

SECONDARY OUTCOMES:
Concentration in plasma of minodronate and alendronate on the first day before administration | on the first day before administration
  Minodronate and alendronate concentration in plasma
Concentration in plasma of minodronate and alendronate on the 8th week after administration | on the 8th week after administration
  Minodronate and alendronate concentration in plasma
Concentration in plasma of minodronate and alendronate on the 12th week after administration | on the 12th week after administration
  Minodronate and alendronate concentration in plasma
Concentration in plasma of minodronate and alendronate on the 24th week after administration | on the 24th week after administration
  Minodronate and alendronate concentration in plasma
Maximum concentration of minodronate and alendronate within 24 weeks | 0-24 weeks
  The observed maximum concentration following administration (Cmax) in plasma after minodronate and alendronate administration.
AUC of minodronate and alendronate within 24 weeks | 0-24 weeks
  The area under the concentration-time curve (AUC) in plasma after minodronate and alendronate administration.
Apparent clearance of minodronate and alendronate within 24 weeks | 0-24 weeks
  The apparent clearance (CL/F) of minodronate and alendronate after administration.
The pharmacodynamic of minodronate and alendronate on the first day before administration | on the first day before administration
  Assessment of bone mineral density at the lumbar spine, and total hip
The pharmacodynamic of minodronate and alendronate on the 12th week after administration | on the12th week after administration
  Assessment of bone mineral density at the lumbar spine, and total hip
The pharmacodynamic of minodronate and alendronate on the 24th week after administration | on the 24th week after administration
  Assessment of bone mineral density at the lumbar spine, and total hip
The incidence of upper gastrointestinal symptoms | 0-24 weeks
  The incidence of upper gastrointestinal symptom after medication administration

CONTACTS AND LOCATIONS:
Overall Officials: Chunli Song, Pro., Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Yoshioka T, Okimoto N, Okamoto K, Sakai A. A comparative study of the effects of daily minodronate and weekly alendronate on upper gastrointestinal symptoms, bone resorption, and back pain in postmenopausal osteoporosis patients. J Bone Miner Metab. 2013 Mar;31(2):153-60. doi: 10.1007/s00774-012-0393-x. Epub 2012 Oct 19. PMID 23076293
- [Derived] Wang H, Huang J, Tao L, Liu D, Song C. Efficacy and safety of minodronate in the treatment of postmenopausal osteoporosis with low back pain: a single-centre, randomized and open-label controlled trial. Trials. 2024 Aug 13;25(1):534. doi: 10.1186/s13063-024-08364-7. PMID 39135126